CLINICAL TRIAL: NCT01957150
Title: Multi-centre, Randomized, Double-blind, Parallel-group Study Evaluating the Effect of Fluticasone Furoate/ Vilanterol (FF/VI) Inhalation Powder Once Daily Compared With Vilanterol (VI) Inhalation Powder Once Daily on Bone Mineral Density (BMD) in Subjects With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Study Evaluating the Effect of Fluticasone Furoate/ Vilanterol (FF/VI) Inhalation Powder Compared With Vilanterol (VI) Inhalation Powder on Bone Mineral Density (BMD) in Subjects With Chronic Obstructive Pulmonary Disease (COPD).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102972; 2012-004801-28 (EudraCT Number)
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate/Vilanterol 100/25 micrograms (mcg) QD (Experimental): Subjects will self administer FF/VI 100/25 mcg inhalation powder once daily for 156 weeks via the NDPI.
  Interventions: Drug: Fluticasone Furoate/Vilanterol
- Vilanterol 25 mcg QD (Experimental): Subjects will self administer VI 25 mcg inhalation powder once daily for 156 weeks via the NDPI.
  Interventions: Drug: Vilanterol

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol — Dry white powder containing 100 mcg of Fluticasone Furoate blended with lactose per blister was administered by NDPI. Dry white powder containing 25 mcg of Vilanterol micronised drug (as the 'M' salt triphenylacetate) blended with lactose and magnesium stearate per blister was administered by NDPI.
  Arms: Fluticasone Furoate/Vilanterol 100/25 micrograms (mcg) QD
Drug: Vilanterol — Dry white powder containing 25 mcg of Vilanterol micronised drug (as the 'M' salt triphenylacetate) blended with lactose and magnesium stearate per blister was administered by NDPI.
  Arms: Vilanterol 25 mcg QD

SUMMARY:
This is a multi-center, randomized, double-blind, parallel-group study. The FF/VI inhalation powder once daily and VI inhalation powder once daily will be evaluated in subjects with COPD over 156 weeks. The primary objective of this study is to evaluate the effect of the inhaled corticosteroid FF on bone mineral density assessed at the total hip by comparing FF/VI treatment with VI treatment in subjects with moderate COPD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Subjects must give their signed and dated written informed consent to participate.
* Gender: Male or female subjects. Female subjects must be post-menopausal or using a highly effective method for avoidance of pregnancy. The decision to include or exclude women of childbearing potential may be made at the discretion of the investigator in accordance with local practice in relation to adequate contraception.
* Age: >= 40 years of age at Screening (Visit 1)
* COPD diagnosis: Subjects with a clinical history of COPD in accordance with the following definition by the American Thoracic Society/European Respiratory Society: COPD is a preventable and treatable disease characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.
* Tobacco use: Subjects with a current or prior history of >=10 pack-years of cigarette smoking at screening (Visit 1). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Number of pack years = (number of cigarettes per day/20) x number of years smoked Note: Pipe and/or cigar use cannot be used to calculate pack year history.
* Severity of Disease: Subject with a measured post-albuterol/salbutamol Forced expiratory volume (FEV1)/forced vital capacity (FVC) ratio of <0.70 at Screening (Visit 1). Subjects with a measured post-albuterol/salbutamol 50% <=FEV1 <=70% of predicted normal values calculated using National Health and Nutrition Examination Survey (NHANES III) reference equations at Screening (Visit 1).
* Native Hip: Have at least one evaluable native hip.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD).
* Alpha1-antitrypsin deficiency: Subjects with alpha-1 antitrypsin deficiency as the underlying cause of COPD.
* Other respiratory disorders: Subjects with tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* Lung resection or transplantation: Subjects with lung volume reduction surgery within the 12 months prior to Screening Visit 1 or having had a lung transplant.
* Chest X-ray: Subjects with a chest X-ray (or Computer Axial Tomography (CT) scan) that revealed evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray should be taken at Screening Visit 1 if a chest X-ray or CT scan is not available within 12 months prior to Visit 1.
* Poorly controlled COPD: Subjects with poorly controlled COPD, defined as the occurrence of the following in the 12 weeks prior to Screening Visit 1: Acute worsening of COPD that is managed by the subject with corticosteroids or antibiotics or that requires treatment prescribed by a physician or requires hospitalization.
* Moderate or severe COPD exacerbation or lower respiratory tract infection: Subjects with 2 or more moderate or severe COPD exacerbations and/or a lower respiratory tract infection (including pneumonia) within the 12 months prior to Screening Visit 1 or experience a moderate or severe COPD exacerbation and/or a lower respiratory infection (including pneumonia) during the Run-In period. NOTE: A moderate COPD exacerbation is defined as requiring systemic corticosteroids and/or antibiotics. A severe COPD exacerbation is defined as requiring hospitalization.
* Abnormal clinically significant laboratory finding: Subjects who have an abnormal, clinically significant finding in any liver chemistry, biochemical, or haematology tests at Screening Visit 1 or upon repeat prior to randomization.
* Abnormal and clinically significant 12-lead Electrocardiogram (ECG): Subjects who have an abnormal, clinically significant ECG finding at Screening Visit 1.
* Non-Compliance during Run-In Period: Failure to demonstrate adequate compliance with run-in medication (< 80% compliant), the ability to withhold COPD medications, and to keep clinic visit appointments.
* Bone disorders/conditions: Subjects with historical or current evidence of bone cancer, severe scoliosis, rheumatoid arthritis, metabolic bone diseases (other than osteoporosis) including hyper-or hypo-parathyroidism, Paget's disease of bone, osteomalacia, or osteogenesis imperfecta. Removal of vertebrae between L1 and L4 of the lumbar spine and/or presence of metal implants or devices, such as plates, rods, or screws in the lumbar spine and/or hip.
* Immobility: Wheel chair bound or paraplegic.
* Low vitamin D: Previously known low-serum 25-hydroxy vitamin D concentration (less than 10ng [25nmoles] per liter).
* Other diseases/abnormalities: Serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study within the 3-year study.
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded if the subject has been considered cured within 5 years since diagnosis.
* Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medications (e.g. beta-agonists, corticosteroid) or components of the inhalation powder (e.g. lactose, magnesium stearate). In addition, patients with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates the subject's participation will also be excluded.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Prohibited medications prior to spirometry at Visit 1: Subjects who are medically unable to withhold the following medications prior to spirometry testing at Visit 1
* No use within 48 hours (hrs) prior to Visit 1 Spirometry Testing: Inhaled corticosteroids, Inhaled Inhaled Corticosteroids (ICS)/ long acting beta2-agonist (LABA) combination products, Long-acting anticholinergics (e.g., tiotropium), Theophylline preparations, Oral leukotriene inhibitors (zafirlukast, montelukast, zileuton), Oral PDE-4 inhibitors (e.g. roflumilast), Oral beta-agonists (Long-acting), Inhaled long acting beta2-agonist (LABA)-Indacaterol.
* No use within 24 hrs prior to Visit 1 Spirometry Testing: Other inhaled LABAs (e.g., salmeterol), Inhaled sodium cromoglycate or nedocromil sodium.
* No use within 12 hrs prior to Visit 1 Spirometry Testing: Oral beta-agonists (Short-acting).
* No use within 4 hrs prior to Visit 1 Spirometry Testing: Ipratropium/ albuterol (salbutamol) combination product, Inhaled short-acting beta2-agonists, Short-acting anti-cholinergics (e.g., ipratropium bromide).
* Additional medication: Use of the following medications within the following time intervals prior to Visit 1 or during the study (unless otherwise specified):
* No use within 12 weeks prior to Screening Visit 1 or thereafter at any time during the study (unless otherwise specified): Depot corticosteroids.
* No use within 30 days prior to Screening Visit 1 or thereafter at any time during the study (unless otherwise specified): Systemic, Oral, parenteral, intra-articular corticosteroids (Subjects may take courses of systemic corticosteroids, where necessary, for treatment of an exacerbation during the double-blind treatment period).
* No use within 30 days or 5 half lives whichever is longer prior to Screening Visit 1 or thereafter at any time during the study (unless otherwise specified): Any other investigational drug.
* COPD medications: Use of ICS, long-acting beta2-agonists (LABA), or ICS/LABA combination products (other than the study-provided double-blind study medication) at Visit 2 (Randomization) or during the double-blind treatment period.
* Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen prn use (i.e., <=12 hours per day) is not exclusionary.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- United States (17):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Old Point Station, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Spokane Valley, Washington
- Canada (5):
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- Germany (6):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Netherlands (8):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Beek
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Losser
  - GSK Investigational Site, Voerendaal
- Spain (8):
  - GSK Investigational Site, Barcelona, Catalonia
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Ponferrada (León)
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Salamanca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted on participants with chronic obstructive pulmonary disease (COPD) in five countries to assess the long-term safety effects of Fluticasone Furoate (FF) component of the FF/Vilanterol (VI) inhalation powder.
Pre-assignment Details: A total of 482 participants were screened of which 199 were screen failures. A total of 283 participants were randomized in a 1:1 ratio to receive either VI or FF/VI.
Groups:
- Participants Administered VI: Following run-in period of 14 to 21 days, eligible participants were administered VI 25 microgram (mcg) once daily via ELLIPTA inhaler for 156 weeks.
- Participants Administered FF/VI: Following run-in period of 14 to 21 days, eligible participants were administered FF 100 mcg along with VI 25 mcg once daily via ELLIPTA inhaler for 156 weeks.
Period: Overall Study
Arm/Group | Participants Administered VI | Participants Administered FF/VI
Started | 142 | 141
Completed | 87 | 83
Not Completed | 55 | 58
Not completed — Adverse Event | 23 | 20
Not completed — Withdrawal by Subject | 13 | 17
Not completed — Physician Decision | 3 | 6
Not completed — Lost to Follow-up | 4 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Administered VI | Participants Administered FF/VI | Total
Number analyzed (Participants) | 142 | 141 | 283
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety population
  Years | 66.0 (8.19) | 64.4 (9.04) | 65.2 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety population
  Participants
    Female | 70 | 71 | 141
    Male | 72 | 70 | 142
Race/Ethnicity, Customized [Number; unit: Count of participants] — Safety population
  Count of participants
    Central/South Asian Heritage | 0 | 1 | 1
    Black or African American | 1 | 1 | 2
    White | 141 | 139 | 280

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Bone Mineral Density (BMD) Measured at Total Hip
Description: BMD analysis performed on log (BMD ratio to baseline) using a repeated measures model with covariates of treatment group, age, gender, baseline BMI, visit, log baseline BMD, log baseline BMD by visit and treatment group by visit interactions. These estimates were then converted into annual changes and averaged to calculate the overall treatment estimates and difference which were used for testing non-inferiority. The analysis shown is for the "While on Treatment" estimand of the difference in percentage change from baseline per annum between FF/VI ± BMD medication/SCS (systemic corticosteroids) and VI ± BMD medication/SCS. Baseline is defined as the measurement performed at Visit 1. Percentage change is calculated as (BMD value post-Baseline divided by Baseline value) -1 multiplied by 100.
Time Frame: Baseline (Visit 1) and 26, 52, 78, 104, 130 and 156 Weeks
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).All randomized participants who received at least one dose of study treatment were included in Safety Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Participants Administered VI | Participants Administered FF/VI
Number analyzed (Participants) | 132 | 130
Percentage change
  Overall % change per year, n = 132, 130 | 0.18 [-0.18 to 0.55] | -0.27 [-0.63 to 0.09]
  % change by Week 26, n= 130, 130: number analyzed (Participants) | 130 | 130
  % change by Week 26, n= 130, 130 | 0.37 [-0.07 to 0.82] | 0.31 [-0.13 to 0.76]
  % change by Week 52, n = 104, 121: number analyzed (Participants) | 104 | 121
  % change by Week 52, n = 104, 121 | 0.35 [-0.21 to 0.91] | -0.43 [-0.96 to 0.10]
  % change by Week 78, n = 97, 102: number analyzed (Participants) | 97 | 102
  % change by Week 78, n = 97, 102 | 0.22 [-0.41 to 0.85] | -0.68 [-1.29 to -0.07]
  % change by Week 104, n = 94, 96: number analyzed (Participants) | 94 | 96
  % change by Week 104, n = 94, 96 | -0.16 [-0.84 to 0.52] | -1.02 [-1.68 to -0.36]
  % change by Week 130, n = 88, 84: number analyzed (Participants) | 88 | 84
  % change by Week 130, n = 88, 84 | 0.00 [-0.73 to 0.75] | -1.02 [-1.75 to -0.29]
  % change by Week 156, n = 76, 75: number analyzed (Participants) | 76 | 75
  % change by Week 156, n = 76, 75 | -0.16 [-1.02 to 0.71] | -1.29 [-2.13 to -0.45]
Statistical Analysis 1: Comparison: Participants Administered VI vs Participants Administered FF/VI; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of 95 % confidence interval (CI) for the overall treatment difference change from Baseline between FF/VI and VI was greater than -1 % year; Percentage Change from Baseline = -0.46, 95% CI 2-sided [-0.97 to 0.06] — Treatment comparison for overall weeks

2. Secondary Outcome: Percentage Change From Baseline in BMD Measurements at Total Hip by Gender (Male Participants)
Description: BMD analysis performed on log (BMD ratio to baseline) using separate repeated measures models for each gender with covariates of treatment group, age, baseline BMI, visit, log baseline BMD, log baseline BMD by visit and treatment group by visit interactions. These estimates were then converted into annual changes and averaged to calculate the overall treatment estimates and difference which were used for testing non-inferiority. The analysis shown is for the "While on Treatment" estimand of the difference in percentage change from baseline per annum between FF/VI ± BMD medication/SCS (systemic corticosteroids) and VI ± BMD medication/SCS. Baseline is defined as the measurement performed at Visit 1. Percentage change is calculated as (BMD value post-Baseline divided by Baseline value) -1 multiplied by 100.
Time Frame: Baseline (Visit 1) and 26, 52, 78, 104, 130 and 156 Weeks
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Participants Administered VI | Participants Administered FF/VI
Number analyzed (Participants) | 67 | 63
Percent change
  Overall Week % change per year, n = 67, 63 | 0.27 [-0.23 to 0.77] | -0.20 [-0.70 to 0.31]
  % change by Week 26, n = 66, 63: number analyzed (Participants) | 66 | 63
  % change by Week 26, n = 66, 63 | 0.45 [-0.06 to 0.97] | 0.44 [-0.09 to 0.97]
  % change by Week 52, n = 52, 56: number analyzed (Participants) | 52 | 56
  % change by Week 52, n = 52, 56 | 0.48 [-0.31 to 1.27] | -0.43 [-1.19 to 0.33]
  % change by Week 78, n = 51, 46: number analyzed (Participants) | 51 | 46
  % change by Week 78, n = 51, 46 | 0.06 [-0.81 to 0.95] | -0.68 [-1.56 to 0.21]
  % change by Week 104, n = 50, 43: number analyzed (Participants) | 50 | 43
  % change by Week 104, n = 50, 43 | 0.07 [-0.86 to 1.00] | -0.68 [-1.62 to 0.27]
  % change by Week 130, n = 44, 39: number analyzed (Participants) | 44 | 39
  % change by Week 130, n = 44, 39 | 0.37 [-0.75 to 1.50] | -0.89 [-2.02 to 0.26]
  % change by Week 156, n = 40, 35: number analyzed (Participants) | 40 | 35
  % change by Week 156, n = 40, 35 | 0.05 [-1.26 to 1.37] | -1.39 [-2.71 to -0.05]
Statistical Analysis 1: Comparison: Participants Administered VI vs Participants Administered FF/VI; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of 95% CI for the overall treatment difference change from Baseline between FF/VI and VI was greater than -1 % year; Percentage Change from Baseline = -0.47, 95% CI 2-sided [-1.17 to 0.24] — Overall Weeks for Male

3. Secondary Outcome: Percentage Change From Baseline in BMD Measurements at Total Hip by Gender (Female Participants)
Description: as for outcome 2
Time Frame: Baseline (Visit 1) and 26, 52, 78, 104, 130 and 156 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Participants Administered VI | Participants Administered FF/VI
Number analyzed (Participants) | 65 | 67
Percent change
  OverallWeek % change per year, n = 65, 67 | 0.09 [-0.46 to 0.64] | -0.31 [-0.84 to 0.22]
  % change by Week 26, n = 64, 67: number analyzed (Participants) | 64 | 67
  % change by Week 26, n = 64, 67 | 0.28 [-0.45 to 1.02] | 0.20 [-0.51 to 0.92]
  % change by Week 52, n = 52, 65: number analyzed (Participants) | 52 | 65
  % change by Week 52, n = 52, 65 | 0.13 [-0.67 to 0.94] | -0.42 [-1.16 to 0.33]
  % change by Week 78, n = 46, 56: number analyzed (Participants) | 46 | 56
  % change by Week 78, n = 46, 56 | 0.37 [-0.54 to 1.28] | -0.63 [-1.48 to 0.23]
  % change by Week 104, n = 44, 53: number analyzed (Participants) | 44 | 53
  % change by Week 104, n = 44, 53 | -0.40 [-1.40 to 0.61] | -1.26 [-2.19 to -0.32]
  % change by Week 130, n = 44, 45: number analyzed (Participants) | 44 | 45
  % change by Week 130, n = 44, 45 | -0.18 [-1.12 to 0.77] | -0.99 [-1.90 to -0.08]
  % change by Week 156, n = 36, 40: number analyzed (Participants) | 36 | 40
  % change by Week 156, n = 36, 40 | -0.42 [-1.56 to 0.73] | -1.19 [-2.27 to -0.11]
Statistical Analysis 1: Comparison: Participants Administered VI vs Participants Administered FF/VI; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Change from Baseline = -0.40, 95% CI 2-sided [-1.16 to 0.36] — Overall Weeks for female

4. Secondary Outcome: Percentage Change From Baseline in BMD Measurements at Lumbar Spine (L1 to L4) by Gender (Male Participants)
Description: as for outcome 2
Time Frame: Baseline (Visit 1) and 26, 52, 78, 104, 130 and 156 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Participants Administered VI | Participants Administered FF/VI
Number analyzed (Participants) | 69 | 64
Percent change
  Overall, male % change per year, n = 69, 64 | 1.41 [0.79 to 2.04] | 0.38 [-0.26 to 1.02]
  % change by Week 26, n = 67, 64: number analyzed (Participants) | 67 | 64
  % change by Week 26, n = 67, 64 | 1.03 [0.26 to 1.80] | 0.42 [-0.36 to 1.21]
  % change by Week 52, n = 53, 56: number analyzed (Participants) | 53 | 56
  % change by Week 52, n = 53, 56 | 1.91 [0.89 to 2.94] | 0.11 [-0.88 to 1.11]
  % change by Week 78, n = 52, 45: number analyzed (Participants) | 52 | 45
  % change by Week 78, n = 52, 45 | 2.09 [0.84 to 3.35] | 0.64 [-0.67 to 1.97]
  % change by Week 104, n = 52, 43: number analyzed (Participants) | 52 | 43
  % change by Week 104, n = 52, 43 | 2.72 [1.48 to 3.98] | 0.42 [-0.88 to 1.75]
  % change by Week 130, n = 47, 38: number analyzed (Participants) | 47 | 38
  % change by Week 130, n = 47, 38 | 1.95 [0.76 to 3.16] | 0.47 [-0.82 to 1.78]
  % change by Week 156, n = 43, 35: number analyzed (Participants) | 43 | 35
  % change by Week 156, n = 43, 35 | 2.96 [1.68 to 4.25] | 1.49 [0.13 to 2.86]
Statistical Analysis 1: Comparison: Participants Administered VI vs Participants Administered FF/VI; Test type: Other; Percentage Change from Baseline = -1.02, 95% CI 2-sided [-1.90 to -0.13] — Overall Weeks for Male

5. Secondary Outcome: Percentage Change From Baseline in BMD Measurements at Lumbar Spine (L1 to L4) by Gender (Female Participants)
Description: as for outcome 2
Time Frame: Baseline (Visit 1) and 26, 52, 78, 104, 130 and 156 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Participants Administered VI | Participants Administered FF/VI
Number analyzed (Participants) | 66 | 68
Percent change
  Overall Week % change per year, n = 66, 68 | 0.17 [-0.42 to 0.77] | 0.12 [-0.45 to 0.70]
  % change by Week 26, n = 66, 68 | 0.10 [-0.67 to 0.88] | -0.19 [-0.95 to 0.58]
  % change by Week 52, n = 51, 66: number analyzed (Participants) | 51 | 66
  % change by Week 52, n = 51, 66 | -0.48 [-1.44 to 0.48] | 0.57 [-0.31 to 1.46]
  % change by Week 78, n = 46, 57: number analyzed (Participants) | 46 | 57
  % change by Week 78, n = 46, 57 | 0.33 [-0.60 to 1.26] | 0.25 [-0.61 to 1.11]
  % change by Week 104, n = 43, 54: number analyzed (Participants) | 43 | 54
  % change by Week 104, n = 43, 54 | 0.65 [-0.50 to 1.80] | 0.64 [-0.41 to 1.70]
  % change by Week 130, n = 44, 49: number analyzed (Participants) | 44 | 49
  % change by Week 130, n = 44, 49 | 1.33 [0.01 to 2.67] | 0.10 [-1.12 to 1.33]
  % change by Week 156, n = 36, 42: number analyzed (Participants) | 36 | 42
  % change by Week 156, n = 36, 42 | 0.80 [-0.74 to 2.36] | 0.10 [-1.32 to 1.53]
Statistical Analysis 1: Comparison: Participants Administered VI vs Participants Administered FF/VI; Test type: Other; Percentage Change from Baseline = -0.05, 95% CI 2-sided [-0.87 to 0.78] — Overall Weeks for female

6. Secondary Outcome: Percentage Change From Baseline in BMD Measurements at Lumbar Spine (L1 to L4)
Description: as for outcome 1
Time Frame: Baseline (Visit 1) and 26, 52, 78, 104, 130 and 156 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Participants Administered VI | Participants Administered FF/VI
Number analyzed (Participants) | 135 | 132
Percentage Change
  Overall week % change per year, n=135, 132 | 0.79 [0.36 to 1.22] | 0.28 [-0.15 to 0.71]
  % change by Week 26, n = 133, 132: number analyzed (Participants) | 133 | 132
  % change by Week 26, n = 133, 132 | 0.55 [0.01 to 1.10] | 0.13 [-0.41 to 0.68]
  % change by Week 52, n = 104, 122: number analyzed (Participants) | 104 | 122
  % change by Week 52, n = 104, 122 | 0.71 [0.01 to 1.42] | 0.40 [-0.26 to 1.07]
  % change by Week 78, n= 98, 102: number analyzed (Participants) | 98 | 102
  % change by Week 78, n= 98, 102 | 1.20 [0.43 to 1.99] | 0.45 [-0.31 to 1.21]
  % change by Week 104, n = 95, 97: number analyzed (Participants) | 95 | 97
  % change by Week 104, n = 95, 97 | 1.66 [0.82 to 2.51] | 0.61 [-0.22 to 1.44]
  % change by Week 130, n = 91, 87: number analyzed (Participants) | 91 | 87
  % change by Week 130, n = 91, 87 | 1.70 [0.80 to 2.61] | 0.30 [-0.60 to 1.20]
  % change by Week 156, n = 79, 77: number analyzed (Participants) | 79 | 77
  % change by Week 156, n = 79, 77 | 1.84 [0.86 to 2.84] | 0.83 [-0.14 to 1.81]
Statistical Analysis 1: Comparison: Participants Administered VI vs Participants Administered FF/VI; Test type: Other; Percentage Change from Baseline = -0.51, 95% CI 2-sided [-1.11 to 0.10] — Overall week

ADVERSE EVENTS:
Time Frame: Serious adverse events and non-serious adverse events were collected from randomization of the study until 159 weeks.
Description: Safety Population. The non-serious AEs are reported using a frequency threshold of >3%.
Arm/Group | Participants Administered VI | Participants Administered FF/VI
All-Cause Mortality (participants affected / at risk) | 6/142 | 4/141
Serious Adverse Events (participants affected / at risk) | 42/142 | 41/141
Other Adverse Events (participants affected / at risk) | 102/142 | 116/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Administered VI (N=142) | Participants Administered FF/VI (N=141)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 6 (10)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 11 (15)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (2) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Administered VI (N=142) | Participants Administered FF/VI (N=141)
Nasopharyngitis (Infections and infestations) | 31 (57) | 40 (75)
Bronchitis (Infections and infestations) | 16 (23) | 11 (12)
Influenza (Infections and infestations) | 5 (5) | 20 (30)
Upper respiratory tract infection (Infections and infestations) | 13 (18) | 12 (20)
Urinary tract infection (Infections and infestations) | 12 (18) | 12 (24)
Sinusitis (Infections and infestations) | 3 (3) | 13 (17)
Pneumonia (Infections and infestations) | 5 (5) | 8 (8)
Oral candidiasis (Infections and infestations) | 4 (5) | 7 (13)
Cystitis (Infections and infestations) | 5 (6) | 5 (7)
Pharyngitis (Infections and infestations) | 4 (5) | 5 (8)
Herpes zoster (Infections and infestations) | 0 (0) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (27) | 20 (28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (13)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (14) | 6 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 13 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 13 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 7 (10)
Constipation (Gastrointestinal disorders) | 3 (4) | 6 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 4 (5)
Toothache (Gastrointestinal disorders) | 3 (3) | 5 (8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 16 (24) | 26 (44)
Hypertension (Vascular disorders) | 11 (12) | 10 (10)
Insomnia (Psychiatric disorders) | 1 (1) | 6 (10)
Anxiety (Psychiatric disorders) | 5 (5) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 6 (7) | 2 (3)
Procedural pain (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (5)
Cataract (Eye disorders) | 3 (3) | 6 (9)
Chest pain (General disorders) | 5 (6) | 4 (4)
Seasonal allergy (Immune system disorders) | 5 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2013-08-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT01957150/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT01957150/SAP_001.pdf